CLINICAL TRIAL: NCT03221881
Title: The Effectiveness and Safety of Neoadjuvant Pegylated Liposomal Doxorubicin and Docetaxel in Breast Cancer.
Brief Title: Neoadjuvant Chemotherapy With a Combination of Pegylated Liposomal Doxorubicin (Caelyx®) and Paclitaxel in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-BC-01
Record Dates: First submitted 2017-06-22; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pegylated Liposomal Doxorubicin and docetaxel (Experimental): Pegylated Liposomal Doxorubicin 30-35 mg/m (2) and docetaxel 75-80 mg/m(2) were both administered on day 1,intravenous, Cycles were repeated in 3-week intervals,for 6 cycles.
  Interventions: Drug: Pegylated Liposomal Doxorubicin and docetaxel

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin and docetaxel
  Other Names: Pegylated Liposomal Doxorubicin 30-35 mg/m (2) and docetaxel 75-80 mg/m(2) were both administered on day 1,intravenous, Cycles were repeated in 3-week intervals,for 6 cycles.

SUMMARY:
In this study, PLD, an anthracycline encapsulated in stealth liposomes, which are believed to efficiently deliver the doxorubicin within the tumour mass with less toxicity compared with standard doxorubicin formulation was used. The study aimed to determine whether the combination of PLD-docetaxel would increase tumour response in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed breast cancer;
2. Age >18 years;
3. Eastern Cooperative Group (ECOG) performance status 0-2;
4. measurable disease (as per radiological imaging); life
5. expectancy >12 months;
6. adequate haematologic blood profile;
7. normal liver and kidney function;
8. adequate cardiac function;
9. no metastatic disease;
10. negative pregnancy test (premenopausal women);
11. signed informed consent.

Exclusion Criteria:

1. Level 2 cardiac toxic effects were deﬁned as asymptomatic systolic dysfunction (NYHA class I) or mildly symptomatic heart failure (NYHA class II) ;
2. Previous treatment for breast cancer, including surgery, radiation, cytotoxic and endocrine treatments (except surgical diagnostic procedures);
3. Active infection or other serious underlying medical or psychiatric condition which would impair the ability of the patient to receive protocol treatment;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
PCR rate | 12 months
  pathologic complete response rate

CONTACTS AND LOCATIONS:
Overall Officials: Shan Baoen, Principal Investigator — Investigator
Locations (1):
- MRI, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No